CLINICAL TRIAL: NCT03830944
Title: Impact of Inflammation-mediated Response on Pan-coronary Plaque Vulnerability, Myocardial Viability and Ventricular Remodeling in the Post-infarction Period - the VIABILITY Study
Brief Title: Inflammation-mediated Coronary Plaque Vulnerability, Myocardial Viability and Ventricular Remodeling
Acronym: VIABILITY
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other); Tîrgu Mureș Emergency Clinical County Hospital, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0119-VIA
Record Dates: First submitted 2019-02-03; First posted 2019-02-05 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2019-07

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: ST elevation myocardial infarction; Inflammatory Response; Coronary plaque vulnerability; myocardial viability
MeSH Terms: conditions — Heart Failure; ST Elevation Myocardial Infarction | interventions — Blood Specimen Collection; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G1: Study subjects with STEMI and increased inflammatory response at 7 days after STEMI
  Interventions:
  * Blood sampling
  * transthoracic echocardiography
  * Late Gadolinium-Enhancement Cardiac Magnetic Resonance
  * Coronary Angio Computed Tomography
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: transthoracic echocardiography; Diagnostic Test: Late Gadolinium-Enhancement Cardiac Magnetic Resonance; Diagnostic Test: Coronary Angio Computed Tomography
- G2: Study subjects with STEMI and no increased inflammatory response at 7 days after STEMI
  Interventions:
  * Blood sampling
  * transthoracic echocardiography
  * Late Gadolinium-Enhancement Cardiac Magnetic Resonance
  * Coronary Angio Computed Tomography
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: transthoracic echocardiography; Diagnostic Test: Late Gadolinium-Enhancement Cardiac Magnetic Resonance; Diagnostic Test: Coronary Angio Computed Tomography

INTERVENTIONS:
Diagnostic Test: Blood sampling — Assessment of complete blood count, biochemistry, inflammatory biomarkers, adhesion molecules
Diagnostic Test: transthoracic echocardiography — Assessment of the ventricular anatomy, size, function, speckle tracking, myocardial strain, valvular function.
Diagnostic Test: Late Gadolinium-Enhancement Cardiac Magnetic Resonance — Assessment of the ventricular anatomy, function, viability, degree of fibrosis, quantification of infarct size, mass.
Diagnostic Test: Coronary Angio Computed Tomography — Assessment of coronary plaque anatomy, morphology, vulnerability features, quantification of epicardial adipose tissue

SUMMARY:
VIABILITY study aims to investigate the link between systemic inflammation, pancoronary plaque vulnerability (referring to the plaque vulnerability within the entire coronary tree), myocardial viability and ventricular remodeling in patients who had suffered a recent ST-segment elevation acute myocardial infarction (STEMI). The level of systemic inflammation in the acute phase of the myocardial infarction and at 1 month will be assessed on the basis of serum levels of inflammatory biomarkers (hsCRP, matrix metalloproteinases, interleukin-6). Pancoronary plaque vulnerability will be assessed: (1) in the acute phase of the infarction, based on serum biomarkers known to be associated with increased plaque vulnerability, such as adhesion molecules (V-CAM or I-CAM) determined from the blood samples collected in the first day after STEMI; (2) at 1 month after infarction, based on computed tomographic angiography analysis of vulnerability features present in all coronary plaques. Myocardial viability and remodeling will be assessed based on: (1) 3D speckle tracking echocardiography associated with dobutamine infusion; (2) MRI imaging associated with complex post-processing techniques for mapping myocardial fibrosis and scar at the level of left atrium and left ventricle. At the same time, CT imaging features associated with systemic and local inflammation, such as global epicardial fat or local pericoronary epicardial fat will be quantified in order to investigate the impact of inflammatory-mediated plaque vulnerability on the extent of myocardial damage in acute myocardial infarction. All these parameters will be investigated in patients with successful primary revascularization performed in a timely manner for ST-segment elevation acute myocardial infarction, who will be divided into 2 groups: group 1 - patients who present persistence of an augmented inflammatory status defined as serum levels of hsCRP>3.0 mg/dl at discharge from the hospital or at 7 days postinfarction (whichever comes first), and group 2 - patients with no persistence of augmented inflammatory status (hsCRP<3.0 mg/dl).

The primary endpoint of the study will be represented by the rate of post-infarction heart failure development, defined as the rate of re-admission in the hospital for heart failure or by a significant decrease in the ejection fraction (<45%).

The secondary endpoints of the study will be:

* rate of re-hospitalization
* rate of repeated revascularization
* rate of major adverse cardiovascular events (MACE rate, including cardiovascular death or stroke)

DETAILED DESCRIPTION:
Patients with acute myocardial infarction (AMI) who survive the acute event, very often present a significant deterioration of their clinical status with progression towards heart failure, which is directly linked to the extent of myocardial injury and the remodeling process starting immediately after infarction. The major aim of the urgent revascularization in STEMI is to save myocardial tissue from death and necrosis, in order to recover viable myocardium. It is well-known that one of the major factors that trigger an AMI is the systemic inflammation, which has a direct influence on coronary plaque vulnerability. At the same time, 20% of patients surviving an AMI present a recurrent cardiovascular event in the following 12 months, as a result of increased systemic inflammation triggered by the infarction, which leads to vulnerabilization of other atheromatous plaques from all the circulatory system in the post-infarction period. While the role of inflammation in acute coronary events is well established, the impact of inflammatory-mediated vulnerability of coronary plaques from the entire coronary tree on the extension of ventricular remodeling and scaring has not been elucidated so far.

This is a clinical prospective, descriptive, single-center study which will be carried out in the University of Medicine, Pharmacy, Science and Technology Tîrgu Mures, Romania, in collaboration with two clinical sites: Center of Advanced Research in Multimodal Cardiac Imaging Cardio Med Tîrgu Mures, Romania and County Clinical Emergency Hospital Tîrgu Mures, Romania. The duration of the study is 2 years which includes the initial screening and the follow-up period.

The study will enroll 100 subjects with STEMI who underwent successful revascularization of the culprit lesion in the first 12 hours after the onset of symptoms. Imaging biomarkers and laboratory analyses such as: high sensitive C Reactive Protein (hsCRP), matrix metalloproteinases (MMP), interleukin-6 (IL6) and N-Terminal Pro-B-Type Natriuretic Peptide (NT pro-BNP) will be determined in the first 24 hours after the index hospitalization. At 1 month postinfarction all patients will undergo Dobutamine stress test associated with speckle tracking echocardiography for evaluation of myocardial function and viability, CMR for assessment of myocardial scar, function and remodeling, and Multislice Angio CT for assessment of pancoronary vulnerability, by complex characterization of vulnerability features in all the coronary plaques present in the coronary tree. All these parameters will be investigated in patients with successful primary percutaneous coronary revascularization, who will be divided into 2 groups: group 1 -patients with persistent elevation of systemic inflammatory biomarkers at discharge from the hospital or at day 7 (whichever comes first) (inflammation+ group); and group 2 - patients with no persistent elevation of systemic inflammatory biomarkers at discharge from the hospital or at day 7 (whichever comes first) (inflammation- group). In all patients, the following biomarkers will be determined: serum levels of inflammatory biomarkers, adhesion molecules and NT-proBNP at 24 hours and 7 days post procedure, the amount of myocardial fibrosis and scar in the left ventricle at 1 month, the degree of ventricular remodeling and myocardial perfusion at 1 month and the amount of epicardial fat surrounding the heart and the plaques. The study will be conducted over a period of 2 years, in which patients will be examined at baseline, and will be followed-up for MACE incidence.

All patients will sign an informed written consent and will be checked for the exclusion criteria prior to enrollment.

Study objectives:

Primary: To investigate the link between coronary inflammation-mediated plaque vulnerability, myocardial viability and ventricular remodeling in the post-infarction period.

Secondary:

* To investigate the impact of systemic inflammation on structural remodeling of the left ventricle in the post-infarction period
* To investigate the impact of local inflammatory response on pancoronary plaque vulnerability following an acute myocardial infarction.

Study Timeline:

* Baseline - visit 1 (day 0)
* Obtain and document consent from participant on study consent form.
* Verify inclusion/exclusion criteria.
* Obtain demographic information, medical history, medication history, alcohol and tobacco use history.
* Record results of physical examinations and 12-lead ECG.
* Collect blood specimens (complete blood count, biochemistry, inflammatory biomarkers, acute adhesion molecules).
* Imaging procedures: transthoracic 2-D echocardiography/speckle tracking
* Visit 2 (day 7 / discharge from the hospital)
* -hsCRP
* Visit 3 (month 1)
* Coronary Computed Tomographic Angiography (vulnerability features, epicardial fat, myocardial perfusion)
* Cardiac Magnetic Resonance (myocardial fibrosis/scar, remodeling, viability)
* Dobutamine stress echocardiography / speckle tracking (viability)
* Visit 4,5,6 (month 3,6,9)
* Record results of physical examinations, 12-lead ECG and medical history.
* Imaging procedures: transthoracic 2-D echocardiography
* Final study visit (month 12)
* Record results of physical examinations, medical history,12-lead ECG
* Imaging procedures: transthoracic 2-D echocardiography
* End-point evaluation.

Study procedures:

* Medical history, clinical examination, laboratory tests (complete blood count, biochemistry, serum level of hs-CRP, MMP, IL6, NT-pro-BNP, adhesion molecules);
* 12-lead ECG
* 2D transthoracic echocardiography with measurement of: cardiac diameters, volumes, left ventricular systolic and diastolic function, speckle tracking echo, dobutamine viability test.
* Late Gadolinium-Enhancement Cardiac Magnetic Resonance (LGE-CMR) with the evaluation of myocardial scar and fibrosis, ventricular function and remodeling index.
* Angio Computed Tomography with assessment of coronary plaque vulnerability (based on vulnerability features: positive remodeling, spotty calcification, napkin-ring sign, low density plaque) and myocardial perfusion Data collection: All the information will be collected in a database that consists of patient's background, medical history, medication, imaging features provided by cardiac ultrasound, Cardiac magnetic resonance, Angio CT and imaging post-processing data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-segment elevation acute myocardial infarction treated by primary PCI within the first 12 hours after the onset of symptoms
* Ability to provide informed consent;
* Patients aged at least 18 years;

Exclusion Criteria:

* Patients with acute coronary syndrome in the last 30 days
* Unwillingness or incapacity to provide informed consent;
* Allergy to contrast media;
* Absolute or relative contraindications to magnetic resonance imaging
* Pregnancy or lactation;
* Women with childbearing potential in absence of any contraceptive treatment
* Renal insufficiency (creatinine greater than 1.5 mg/dL) or renal failure requiring dialysis;
* Active malignancy or malignancy within the last 5 year prior to enrollment;
* Conditions associated with an estimated life expectancy of under 1 year;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients from a single center with STEMI meeting inclusion and exclusion criteria and undergoing primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of post-infarction heart failure | 12 months
  The primary outcome measure will be represented by the rate of post-infarction heart failure development, defined as the rate of re-admission in the hospital for heart failure or by a significant decrease in the ejection fraction (<45%).

SECONDARY OUTCOMES:
Rate of re-hospitalization | 12 months
  Re-hospitalization for cardiovascular related causes
Rate of repeated revascularization | 12 months
  Repeated myocardial revascularization procedures
Rate of major adverse cardiovascular events | 12 months
  Occurrence of major adverse cardiovascular events described as cardiovascular death, stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Mirabela Morariu, MD, Principal Investigator — University of Medicine, Pharmacy, Science and Technology of Tîrgu Mures, Romania
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD sharing frame is starting 6 months after publication.